CLINICAL TRIAL: NCT01604941
Title: A Phase 2, 24 Week, Open Label, Multi-Center Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SSP-004184 (SPD602) in the Treatment of Chronic Iron Overload Requiring Chelation Therapy
Brief Title: Pharmacokinetics of SSP-004184 in the Treatment of Chronic Iron Overload Requiring Chelation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to treatment stop resulting in an inability to draw conclusions from the data. Evaluation of nonclinical rat findings is ongoing.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD602-203; FBS0701-CTP-16 (Other: Ferrokin); 2011-005675-16 (EudraCT Number)
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Iron Overload Due to Repeated Red Blood Cell Transfusions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SPD602 (Experimental): 50 mg/kg/day orally twice daily for 24 weeks
  Interventions: Drug: SPD602

INTERVENTIONS:
Drug: SPD602 — 50 mg/kg/day orally twice daily for 24 weeks
  Other Names: SSP-004184, deferitazole

SUMMARY:
The purpose of this study is to evaluate SSP-004184AQ in patients with transfusional iron overload whose primary diagnosis is hereditary or congenital anemia.

SSP-004184AQ is an iron chelator under development for chronic daily oral administration to patients with transfusional iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign the approved informed consent.
* Age: 18-60 years old, inclusive, at Screening.
* Subjects who have received more than 20 transfusions in their lifetime and who have transfusional iron overload requiring chronic treatment with an iron chelator. N.B.: Sickle Cell Disease subjects receiving regular exchange transfusions and iron overloaded subjects with thalassemia intermedia who are receiving regular transfusions (transfusion dependent thalassemia intermedia) are eligible.
* Willing to discontinue all existing iron chelation therapies for a minimum period of one to five days prior to first dose of SSP-004184AQ, the 24 week duration of the study and 1 week after last dose for a total of approximately 26 weeks.
* Willing to fast two hours prior to and one hour after each dose.
* Serum ferritin >500ng/mL at Screening.
* Baseline liver iron concentration is greater than or equal to 5mg iron per g (equivalent dry weight, liver)determined by FerriScan® R2 MRI.
* Mean of the previous three pre-transfusion hemoglobin concentrations is greater than or equal to 7.5g/dL.
* Adult female subjects should be:

  1. Post-menopausal (12 consecutive months of spontaneous amenorrhea), or
  2. Surgically sterile, or
  3. Females of child-bearing potential must have a negative beta-HCG pregnancy test at the Screening Visit and a negative urine pregnancy test at the Baseline Visit.

Females of child-bearing potential must agree to abstain from sexual activity that could result in pregnancy or agree to use acceptable methods of contraception.

Exclusion Criteria:

* As a result of medical review, physical examination, or Screening investigations, the Principal Investigator (PI) considers the subject unfit for the study.
* Non-elective hospitalization within the 30 days prior to Baseline testing.
* Evidence of clinically relevant oral, cardiovascular, gastrointestinal, hepatic, biliary, renal, endocrine, pulmonary, neurologic, psychiatric, immunologic, bone marrow, or skin disorder that contraindicates dosing with SSP-004184AQ.
* Iron overload from causes other than transfusional siderosis.
* Evidence of severe renal insufficiency, eg, serum creatinine 1.5X above the upper limit of normal or proteinuria greater than 1 gm per day or a calculated glomerular filtration rate <60mL/min.
* Severe iron overload including:

  1. T2* MRI <10 ms
  2. liver iron concentration by FerriScan R2 MRI >30mg/g liver (dw)
* Known sensitivity to magnesium stearate, croscarmellose sodium or SSP-004184AQ.
* Platelet count below 100,000/μL or absolute neutrophil count less than 1500/mm3 at Screening.
* Insufficient venous access that precludes prescribed blood draws for safety laboratory assessments.
* ALT at Screening >200 IU/L.
* Use of any investigational agent within the 30 days prior to the Baseline testing.
* Pregnant or lactating females.
* Cardiac left ventricular ejection fraction

  1. Below the locally determined normal range in the 12 months prior to Screening by echocardiograph or MRI or
  2. <50% at Baseline testing by MRI (echocardiograph is acceptable for LVEF if MRI information is not available).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-09-14 (Actual); Primary Completion 2014-04-18 (Actual); Study Completion 2014-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- United States (4):
  - Children's Center for Cancer and Blood Diseases, Los Angeles, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Weill Cornell Medical College, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Toronto General Hospital, Toronto, Ontario, Canada
- Egypt (2):
  - Ain Shams University Pediatric Hospitals, Cairo
  - Cairo University Pediatric Hospitals, Cairo
- Italy (4):
  - Centro della Microcitemia e delle Anemie Congenite, Genova, Genoa
  - San Luigi Hospital Thalassemia Centre, Orbassano, Torino
  - Ospedale Regionale Microcitemie, Cagliari
  - Ospedale Maggiore Policlinico, Milan
- American University of Beirut Medical Center, Beirut, Lebanon

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study started as a double-arm study with once daily (QD) dosing but was amended first to a double-arm study with twice daily (BID) dosing and then to a single-arm study after removing the higher dose. Some participants were enrolled directly to BID dosing, some to QD dosing and then re-enrolled to BID dosing, some completed with QD dosing.
Groups:
- SPD602 50mg/mg/Day Twice Daily Dosing (BID): Participants were randomly assigned to 50 mg/kg/day oral BID dosing and continued BID dosing until the end of study (24 weeks) or early discontinuation.
- SPD602 75mg/kg/Day Twice Daily Dosing (BID): Participants were randomly assigned to 75 mg/kg/day oral BID dosing and continued BID dosing until the end of study (24 weeks) or early discontinuation.
- SPD602 50mg/kg/Day Once (QD) Then Twice Daily Dosing (BID): Participants were randomly assigned to QD dosing then re-enrolled to 50 mg/kg/day oral BID dosing and continued BID dosing until the end of study (24 weeks) or early discontinuation.
- SPD602 75mg/kg/Day Once (QD) Then Twice Daily Dosing (BID): Participants were randomly assigned to QD dosing then re-enrolled to 75 mg/kg/day oral BID dosing and continued BID dosing until the end of study (24 weeks) or early discontinuation.
- SPD602 50mg/kg/Day Once Daily Dosing (QD): Participants were randomly assigned to 50 mg/kg/day oral QD dosing and continued QD dosing until the end of study (24 weeks) or early discontinuation.
- SPD602 75mg/kg/Day Once Daily Dosing (QD): Participants were randomly assigned to 75 mg/kg/day oral QD dosing and continued QD dosing until the end of study (24 weeks) or early discontinuation.
Period: Overall Study
Arm/Group | SPD602 50mg/mg/Day Twice Daily Dosing (BID) | SPD602 75mg/kg/Day Twice Daily Dosing (BID) | SPD602 50mg/kg/Day Once (QD) Then Twice Daily Dosing (BID) | SPD602 75mg/kg/Day Once (QD) Then Twice Daily Dosing (BID) | SPD602 50mg/kg/Day Once Daily Dosing (QD) | SPD602 75mg/kg/Day Once Daily Dosing (QD)
Started | 11 | 4 | 3 | 3 | 4 | 7
Completed | 0 | 0 | 0 | 0 | 3 | 0
Not Completed | 11 | 4 | 3 | 3 | 1 | 7
Not completed — Adverse Event | 1 | 2 | 0 | 0 | 1 | 5
Not completed — Non-compliance | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Decision | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Early Study Termination | 9 | 2 | 3 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set, defined as all participants who had taken at least 1 BID dose of investigational product.
Groups:
- SPD602 50mg/kg/Day: Participants received SPD602 50mg/kg/day oral dosing either twice daily (BID) or once daily (QD), then BID.
- SPD602 75mg/kg/Day: Participants received SPD602 75mg/kg/day oral dosing either twice daily (BID) or once daily (QD), then BID.
- Total: Total of all reporting groups
Arm/Group | SPD602 50mg/kg/Day | SPD602 75mg/kg/Day | Total
Number analyzed (Participants) | 12 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (5.79) | 24.4 (5.80) | 26.8 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Liver Iron Concentration (LIC) as Assessed by FerriScan R2 Magnetic Resonance Imaging (MRI)
Description: The efficacy of SPD602 was assessed by determining LIC. Abdominal MRI data were collected by using FerriScan R2 standard procedures and used to determine LIC. A negative change from baseline indicates that LIC decreased. Early Termination was within the protocol defined visit date +/- 14 days window and was mapped to next scheduled MRI visit for 3 participants.
Time Frame: Baseline, 12 and 24 weeks
Population: The Full Analysis Set, defined as all participants in the Safety Set who had at least 1 post-baseline primary efficacy assessment. The Safety Set was defined as all participants who had taken at least 1 BID dose of investigational product.
Measure: Mean (Standard Deviation); unit: mg Fe/g*dw
Groups:
- SPD602 50 mg/kg/d: Participants received SPD602 50mg/kg/day oral dosing either twice daily (BID) or once daily (QD), then BID.
- All Participants With BID Dosing: Of the 21 participants randomly assigned to BID dosing (including re-enrolled participants), 10 were excluded from the Full Analysis Set. Data for this arm were analyzed to verify that the protocol, as finally amended, was not impacted by using only the lower dose.
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
mg Fe/g*dw
  Week 12, n=5,10 | -3.4 (6.4) | -3.8 (5.0)
  Week 24, n=1,2 | -5.3 (NA) — Only 1 participant was analyzed | -2.1 (4.5)
Statistical Analysis 1: Comparison: SPD602 50 mg/kg/d; Analysis of Week 12 for 50 mg/kg/d dosing; Test type: Superiority or Other; p = 0.2960, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline
Statistical Analysis 2: Comparison: All Participants With BID Dosing; Analysis of Week 12 for all participants with BID dosing; Test type: Superiority or Other; p = 0.0400, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline
Statistical Analysis 3: Comparison: All Participants With BID Dosing; Analysis of Week 24 for all participants with BID dosing; Test type: Superiority or Other; p = 0.6303, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline

2. Secondary Outcome: Change From Baseline in LIC as Assessed by R2* MRI
Description: The efficacy of SPD602 was assessed by determining LIC. Abdominal MRI data were collected by using R2* standard procedures (liver and pancreas) and used to determine LIC. A negative change from baseline indicates that LIC decreased. Early Termination was within the protocol defined visit date +/- 14 days window and was mapped to next scheduled MRI visit for 3 participants.
Time Frame: Baseline, 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg Fe/g*dw
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
mg Fe/g*dw
  Week 12, n=5,9 | -3.2 (2.3) | -3.2 (2.1)
  Week 24, n=1,2 | -2.4 (NA) — Only 1 participant was analyzed | -3.3 (1.3)
Statistical Analysis 1: Comparison: SPD602 50 mg/kg/d; Analysis of Week 12 for 50 mg/kg/d dosing; Test type: Superiority or Other; p = 0.0365, paired t-test — P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline
Statistical Analysis 2: Comparison: All Participants With BID Dosing; Analysis of Week 12 for all participants with BID dosing; Test type: Superiority or Other; p = 0.0019, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline
Statistical Analysis 3: Comparison: All Participants With BID Dosing; Analysis of Week 24 for all participants with BID dosing; Test type: Superiority or Other; p = 0.1695, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline

3. Secondary Outcome: Change From Baseline in LIC Adjusted by Transfusional Iron Intake And Assessed by R2* MRI
Description: The efficacy of SPD602 was assessed by determining LIC and adjusting for transfusional iron intake. Abdominal MRI data were collected by using R2* standard procedures (liver and pancreas) and used to determine LIC. A negative change from baseline indicates that LIC decreased. For participants who had a blood transfusion on the MRI exam date, the blood transfusion done immediately prior to the MRI exam date was included in the calculation of daily transfusion intake. Early Termination was within the protocol defined visit date +/- 14 days window and was mapped to next scheduled MRI visit for 3 participants.
Time Frame: Baseline, 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg Fe/g*dw
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
mg Fe/g*dw
  Week 12, n=5,9 | -6.0 (4.5) | -6.2 (3.2)
  Week 24, n=1,2 | -9.9 (NA) — Only 1 participant was analyzed | -10.5 (0.8)
Statistical Analysis 1: Comparison: SPD602 50 mg/kg/d; Analysis of Week 12 for 50 mg/kg/d dosing; Test type: Superiority or Other; p = 0.0394, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline
Statistical Analysis 2: Comparison: All Participants With BID Dosing; Analysis of Week 12 for all participants with BID dosing; Test type: Superiority or Other; p = 0.0004, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline
Statistical Analysis 3: Comparison: All Participants With BID Dosing; Analysis of Week 24 for all participants with BID dosing; Test type: Superiority or Other; p = 0.0332, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline

4. Secondary Outcome: Change From Baseline in Cardiac T2* Relaxation Rate, an MRI Parameter Used to Estimate Cardiac Iron Load
Description: The efficacy of SPD602 was assessed by estimating cardiac iron load. T2* data from cardiac MRI were collected by using standard procedures and used as an estimate of cardiac iron load. T2* is an MR relaxation parameter that is reported in milliseconds. Iron within a tissue decreases homogeneity of the magnetic field and shortens the T2* relaxation rate (Anderson, 2001). Low cardiac T2* values are associated with increased risk of heart failure (Kirk, 2009). A negative change from baseline in the T2* relaxation rate indicates that iron load increased. Early Termination was within the protocol defined visit date +/- 14 days window and was mapped to next scheduled MRI visit for 3 participants.
Time Frame: Baseline, 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
milliseconds
  Week 12, n=5,7 | -0.64 (3.080) | -0.24 (3.910)
  Week 24, n=1,2 | -4.10 (NA) — Only 1 participant was analyzed | -2.60 (2.121)
Statistical Analysis 1: Comparison: SPD602 50 mg/kg/d; Analysis of Week 12 for 50 mg/kg/d dosing; Test type: Superiority or Other; p = 0.3202, paired t-test — The P-value is from Paired t-test for log-transformed data at post treatment timepoint vs. Baseline
Statistical Analysis 2: Comparison: All Participants With BID Dosing; Analysis of Week 12 for all participants with BID dosing; Test type: Superiority or Other; p = 0.4549, paired t-test — The P-value is from Paired t-test for log-transformed data at post treatment timepoint vs. Baseline
Statistical Analysis 3: Comparison: All Participants With BID Dosing; Analysis of Week 24 for all participants with BID dosing; Test type: Superiority or Other; p = 0.3291, paired t-test — The P-value is from Paired t-test for log-transformed data at post treatment timepoint vs. Baseline

5. Secondary Outcome: Change From Baseline in Serum Ferritin
Description: Serum ferritin levels were determined from serum biochemistry analyses. A negative change from baseline indicates that serum ferritin decreased.
Time Frame: Baseline, 8 and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
ng/mL
  Week 8, n=5,11 | -762.63 (2100.683) | -568.08 (1426.687)
  Week 16, n=1,4 | 586.47 (NA) — Only 1 participant was analyzed | 137.63 (972.970)
Statistical Analysis 1: Comparison: SPD602 50 mg/kg/d; Analysis of Week 8 for 50 mg/kg/d dosing; Test type: Superiority or Other; p = 0.6703, paired t-test — The P-value is from Paired t-test for log-transformed data at post treatment timepoint vs. Baseline
Statistical Analysis 2: Comparison: All Participants With BID Dosing; Analysis of Week 8 for all participants with BID dosing; Test type: Superiority or Other; p = 0.2618, paired t-test — The P-value is from Paired t-test for log-transformed data at post treatment timepoint vs. Baseline
Statistical Analysis 3: Comparison: All Participants With BID Dosing; Analysis of Week 16 for all participants with BID dosing; Test type: Superiority or Other; p = 0.7679, paired t-test — The P-value is from Paired t-test for log-transformed data at post treatment timepoint vs. Baseline

6. Primary Outcome: Change From Baseline in LIC Adjusted by Transfusional Iron Intake And Assessed by FerriScan R2 MRI
Description: The efficacy of SPD602 was assessed by determining LIC and adjusting for transfusional iron intake. Abdominal MRI data were collected by using FerriScan R2 standard procedures and used to determine LIC. A negative change from baseline indicates that LIC decreased. For participants who had a blood transfusion on the MRI exam date, the blood transfusion done immediately prior to the MRI exam date was included in the calculation of daily transfusion intake. Early Termination was within the protocol defined visit date +/- 14 days window and was mapped to next scheduled MRI visit for 3 participants.
Time Frame: Baseline, 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg Fe/g*dw
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
mg Fe/g*dw
  Week 12, n=5,10 | -6.3 (8.4) | -6.6 (6.7)
  Week 24, n=1,2 | -12.8 (NA) — Only 1 participant was analyzed | -9.3 (5.0)
Statistical Analysis 1: Comparison: SPD602 50 mg/kg/d; Analysis of Week 12 for 50 mg/kg/d dosing; Test type: Superiority or Other; p = 0.1683, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline
Statistical Analysis 2: Comparison: All Participants With BID Dosing; Analysis of Week 12 for all participants with BID dosing; Test type: Superiority or Other; p = 0.0123, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline
Statistical Analysis 3: Comparison: All Participants With BID Dosing; Analysis of Week 24 for all participants with BID dosing; Test type: Superiority or Other; p = 0.2334, paired t-test — The P-value is from analysis of paired t-test at post treatment timepoint vs. Baseline

7. Secondary Outcome: Number of Participants Classified as a Responder by FerriScan R2 MRI Analysis of LIC
Description: A responder was defined as a participant whose observed liver iron concentration (LIC) at the measured time point was less than the baseline value. LIC was assessed by abdominal MRI with the FerriScan R2 according to standard procedures. Early Termination was within the protocol defined visit date +/- 14 days window and was mapped to next scheduled MRI visit for 3 participants.
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
participants
  Week 12, n=5,10 | 4 | 8
  Week 24, n=1,2 | 1 | 1

8. Secondary Outcome: Number of Participants Classified as a Responder by FerriScan R2 MRI Analysis of LIC Adjusted For Transfusional Iron Intake
Description: A responder was defined as a participant whose observed liver iron concentration (LIC) at the measured time point was less than the baseline value. LIC was assessed by abdominal MRI with the FerriScan R2 according to standard procedures, and the results were adjusted for transfusional iron intake. Early Termination was within the protocol defined visit date +/- 14 days window and was mapped to next scheduled MRI visit for 3 participants. For participants who had a blood transfusion on the MRI exam date, the blood transfusion done immediately prior to the MRI exam date was included in the calculation of daily transfusion intake.
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
participants
  Week 12, n=5,10 | 4 | 8
  Week 24, n=1,2 | 1 | 1

9. Secondary Outcome: Number of Participants Classified as a Responder by R2* MRI Analysis of LIC
Description: A responder was defined as a participant whose observed liver iron concentration (LIC) at the measured time point was less than the baseline value. LIC was assessed by abdominal MRI with the R2* according to standard procedures (liver and pancreas). Early Termination was within the protocol defined visit date +/- 14 days window and was mapped to next scheduled MRI visit for 3 participants.
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
participants
  Week 12, n=5,9 | 5 | 9
  Week 24, n=1,2 | 1 | 2

10. Secondary Outcome: Number of Participants Classified as a Responder by R2* MRI Analysis of LIC Adjusted For Transfusional Iron Intake
Description: A responder was defined as a participant whose observed liver iron concentration (LIC) at the measured time point was less than the baseline value. LIC was assessed by abdominal MRI with the R2* according to standard procedures (liver and pancreas), and the results were adjusted for transfusional iron intake. Early Termination was within the protocol defined visit date +/- 14 days window and was mapped to next scheduled MRI visit for 3 participants. For participants who had a blood transfusion on the MRI exam date, the blood transfusion done immediately prior to the MRI exam date was included in the calculation of daily transfusion intake.
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
participants
  Week 12, n=5,9 | 5 | 9
  Week 24, n=1,2 | 1 | 2

11. Secondary Outcome: Number of Participants Classified as a Responder by Serum Ferritin
Description: A responder was defined as a participant whose observed serum ferritin level at the measured time point was less than the baseline value. Serum ferritin levels were determined from serum biochemistry analyses.
Time Frame: 8 and 16 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SPD602 50 mg/kg/d | All Participants With BID Dosing
Number analyzed (Participants) | 5 | 11
participants
  Week 8, n=5,11 | 3 | 8
  Week 16, n=1,4 | 0 | 1

ADVERSE EVENTS:
Description: All safety analyses, including analyses of AEs, were based on the Safety Set, which included participants in the 50mg/kg/day BID and 75mg/kg/day BID dosing groups who had taken at least 1 BID dose of investigational product. Participants in the QD only dosing groups were not included in the Safety Set.
Groups:
- SPD602 50mg/kg/Day: Participants received SPD602 50mg/kg/day oral dosing BID either as originally randomized or as a re-enrolled participant.
- SPD602 75mg/kg/Day: Participants received SPD602 75mg/kg/day oral dosing BID either as originally randomized or as a re-enrolled participant.
Arm/Group | SPD602 50mg/kg/Day | SPD602 75mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 2/12 | 2/7
Other Adverse Events (participants affected / at risk) | 9/12 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD602 50mg/kg/Day (N=12) | SPD602 75mg/kg/Day (N=7)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD602 50mg/kg/Day (N=12) | SPD602 75mg/kg/Day (N=7)
Paraesthesia (Nervous system disorders) | 2 (3) | 4 (5)
Chromaturia (Renal and urinary disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 2 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (4) | 2 (3)
Pyrexia (General disorders) | 3 (7) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (8) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anion gap increased (Investigations) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nitrite urine present (Investigations) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urine protein/creatinine ratio increased (Investigations) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Axillary pain (General disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1)
pH urine increased (Investigations) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 (0) | 1 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated due to treatment stop resulting in an inability to draw conclusions from the data. Evaluation of nonclinical rat findings is ongoing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.